CLINICAL TRIAL: NCT07376512
Title: Predicting Response to Anti-PD-1/PD-L1 Immunotherapy by Plasma Extracellular Vesicle Analysis
Acronym: EVpredict
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-A01783-46
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer; Melanoma (Skin Cancer)
Keywords: standard treatment with anti-PD-(L)1 monotherapy or combination therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Advanced NSCLC or Melanoma - Anti-PD-(L)1 Therapy: This cohort includes patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) or inoperable melanoma who are receiving standard-of-care anti-PD-1 or anti-PD-L1 therapy, either as monotherapy or in combination with other approved therapies.
  Participants will follow standard clinical management, and study-specific procedures include four blood draws for extracellular vesicle (EV) analysis at baseline and during follow-up, collection of standard immunohistochemistry results (PD-1, PD-L1, CTLA-4, Tim-3, LAG-3, TIGIT), thoraco-abdominopelvic CT imaging, and tumor DNA genotyping performed as part of routine care.

SUMMARY:
The objective of this prospective multicenter study is to evaluate whether the analysis of immunological biomarkers present in circulating extracellular vesicles is associated with the response to anti-PD-1/PD-L1 treatments in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) or unresectable melanoma.

Patients will receive standard-of-care treatment and will be followed according to routine clinical practice. The study involves the collection of four study-specific blood samples at different time points during follow-up, as well as the collection of standard immunohistochemistry results, thoraco-abdomino-pelvic CT scans, and tumor DNA genotyping analyses performed as part of routine care.

The study aims to determine:

* whether baseline biomarkers in extracellular vesicles are associated with response to anti-PD-1/PD-L1 treatment,
* how these biomarkers change over the course of treatment, and
* to provide exploratory data for the development of predictive immunological response signatures.

DETAILED DESCRIPTION:
Immune checkpoint inhibitors (anti-PD-1/PD-L1) have become standard treatment for patients with advanced or metastatic non-small cell lung cancer (NSCLC) or melanoma. However, not all patients respond to these therapies, and current biomarkers are imperfect.

Circulating extracellular vesicles (EVs) are nanovesicles derived from tumor and immune cells, carrying proteins, nucleic acids, and lipids. They represent an accessible and stable source of immunological biomarkers, allowing monitoring of the tumor microenvironment without additional invasive procedures.

This prospective multicenter study aims to:

* Collect and analyze immunological biomarkers present in EVs at baseline and during follow-up.
* Assess their association with objective response to anti-PD-1/PD-L1 treatment, measured according to RECIST 1.1.
* Develop an exploratory composite score combining multiple markers to predict response, stratified by cancer type (NSCLC vs melanoma).
* Prospectively collect biological samples for future exploratory analyses.

Study procedures for participants include:

* Blood sample collection: Four study-specific blood draws performed during standard treatment or tumor assessment visits (baseline, 2nd administration, first evaluation, second evaluation).
* Collection of additional information: Standard immunohistochemistry results for PD-1, PD-L1, CTLA-4, Tim-3, LAG-3, and Tigit; thoraco-abdomino-pelvic CT scans; circulating or tumor DNA genotyping analyses.
* Clinical follow-up: Conducted according to routine care standards, with no changes to treatment or additional study-specific visits.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Histologically confirmed diagnosis of non-small cell lung cancer (NSCLC) or locally advanced/metastatic unresectable melanoma.
* Patient scheduled to initiate anti-PD-(L)1 therapy, either as monotherapy or in combination (other immune checkpoint inhibitors, chemotherapy, etc.).
* Baseline tumor assessment performed within 28 days prior to enrollment (CT scan of thorax, abdomen, and pelvis) with at least one measurable lesion according to RECIST 1.1 criteria.
* Life expectancy >6 months.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 at enrollment.
* Patient able to provide informed consent and comply with study procedures.
* Patient covered by a social security system or equivalent.

Exclusion Criteria:

* Prior treatment with immunotherapy.
* Presence of EGFR or ALK mutation (applicable only to the lung cohort).
* Presence of another synchronous malignancy.
* Diagnosis of uveal melanoma.
* Treatment with systemic immunosuppressants, including within 28 days prior to enrollment, or corticosteroids >10 mg/day, including within 14 days prior to enrollment.
* Disease not measurable according to RECIST 1.1 criteria.
* Positive serology for HIV, HBV, or HCV.
* Pregnant or breastfeeding women.
* Inability to comply with study follow-up and visits for geographic, social, or psychological reasons.
* Individuals deprived of liberty or under legal guardianship (including curatorship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-small cell lung cancer (NSCLC) or melanoma, locally advanced or metastatic, and unresectable. For all patients, first-line standard treatment will be based on standard care with an anti-PD-(L)1 therapy, either as monotherapy or in combination (with other immune checkpoint inhibitors or chemotherapy). Standard treatments are defined by the approved indications (marketing authorizations) in France.
Sampling Method: Non-Probability Sample
Enrollment: 378 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Target protein levels in plasma-derived extracellular vesicles (EVs) measured by multiplex ELISA before treatment | 6 months from treatment initiation
  Treatment response assessed as Best Overall Response (BOR: complete or partial response per RECIST 1.1) within 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica JG GOBBO, Clinical Research Scientist, Study Chair — Centre Georges François Leclerc
Locations (5):
- France (5):
  - CHU Besançon - Service Dermatologie, Besançon
  - CHU Besançon - Service Pneumologie Oncologie Thoracique, Besançon
  - Centre Georges-François Leclerc, Dijon
  - CHU Dijon - Service Oncologie Médicale, Dijon
  - Centre Leon Berard - Service Oncologie Médicale, Lyon

IPD SHARING:
Plan to Share IPD: No